CLINICAL TRIAL: NCT00722046
Title: A PHASE 2 MULTICENTER, RANDOMIZED, DOUBLE BLIND, PLACEBO CONTROLLED STUDY OF THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF MULTIPLE DOSES OF PF 04360365 IN PATIENTS WITH MILD TO MODERATE ALZHEIMER'S DISEASE.
Brief Title: Multiple IV Dose Study Of PF-04360365 In Patients With Mild To Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9951002; 2008-000986-42 (EudraCT Number); MD IN AD PATIENT (Other: Alias Study Number)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; antibody; amyloid
MeSH Terms: conditions — Alzheimer Disease | interventions — ponezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- PF-04360365 0.1 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 0.1 mg/kg
- PF-04360365 0.5 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 0.5 mg/kg
- PF-04360365 1 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 1 mg/kg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-04360365 3 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 3 mg/kg
- PF-04360365 8.5 mg/kg (Experimental)
  Interventions: Biological: PF-04360365 8.5 mg/kg

INTERVENTIONS:
Biological: PF-04360365 0.1 mg/kg — 0.1 mg/kg every 60 days (10 doses total)
  Arms: PF-04360365 0.1 mg/kg
Biological: PF-04360365 0.5 mg/kg — 0.5 mg/kg every 60 days (10 doses total)
  Arms: PF-04360365 0.5 mg/kg
Biological: PF-04360365 1 mg/kg — 1 mg/kg every 60 days (10 doses total)
  Arms: PF-04360365 1 mg/kg
Drug: Placebo — Placebo every 60 days (10 doses total)
  Arms: Placebo
Biological: PF-04360365 3 mg/kg — 3 mg/kg every 60 days (10 doses total)
  Arms: PF-04360365 3 mg/kg
Biological: PF-04360365 8.5 mg/kg — 8.5 mg/kg every 60 days (10 doses total)
  Arms: PF-04360365 8.5 mg/kg

SUMMARY:
Purpose of the study is to determine whether multiple dose administration of PF-04360365 is safe and well tolerated in patient with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non childbearing potential, age > or = 50
* Diagnosis of probable Alzheimer's disease, consistent with criterial from both:

  * National Institute of Neurological and Communicable Disease and Stroke and Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
  * Diagnostic and Statistical Manual of Mental Disorders (DSM IV)
* Mini-mental status exam score of 16-26 inclusive
* Rosen-Modified Hachinski Ischemia Score of < or = 4

Exclusion Criteria:

* Diagnosis or history of other demential or neurodegenerative disorders
* Diagnosis or history of clinically significant cerebrovascular disease
* Specific findings on magnetic resonance imaging (MRI); cortical infarct, micro hemorrhage, multiple white matter lacunes, extensive white matter abnormalities
* History of autoimmune disorders
* History of allergic or anaphylactic reactions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-12-05 (Actual); Primary Completion 2011-08-16 (Actual); Study Completion 2011-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (14):
  - Pivotal Research Center, Peoria, Arizona
  - Sun Radiology- for MRI, Peoria, Arizona
  - Dedicated Phase 1, Phoenix, Arizona
  - Neuroscience Consultants, LLC, Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - MRA Clinical Research, South Miami, Florida
  - Sleep Florida, LLC, South Miami, Florida
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Alexian Brothers Neurosciences Institute, Elk Grove Village, Illinois
  - Stark Pharmacy, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Memory Enhancement Center of America, Inc, Eatontown, New Jersey
  - Central Jersey Radiology, Oakhurst, New Jersey
  - Butler Hospital, Providence, Rhode Island
- Australia (4):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital and Health Service, Woodville South, South Australia
  - Heidelberg Repatriation Hospital, Austin Health, Heidelberg West, Victoria
  - The McCusker Foundation for Alzheimer's Disease Research, Nedlands, Western Australia
- Belgium (4):
  - ZNA Middelheim / Neurology, Antwerp
  - UZ Antwerpen, Department of Neurology, Edegem
  - UZ Brussel / Geriatrie, Jette
  - U.Z. Gasthuisberg / Neurologie, Leuven
- Canada (7):
  - University of British Columbia Hospital, Division of Neurology, Vancouver, British Columbia
  - Parkwood Hospital, Geriatric Medicine, London, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Recherche Clinique de Neurologie, Montreal, Quebec
  - Diex Recherche Inc., Sherbrooke, Quebec
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Hanyang University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
- United Kingdom (6):
  - The Pharmacy Department, Cheadle, Chesire
  - The Shalbourne Suite, Swindon, Wiltshire
  - Kingshill Research Centre, Swindon, Wiltshire
  - MAC UK Neuroscience Ltd, Manchester
  - Wellcome Trust Clinical Research Facility, Southampton
  - Memory Assessment and Research Centre, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04360365 0.1 mg/kg (Part A): PF-04360365 0.1 milligram per kilogram (mg/kg) intravenous infusion over 2 hours every 60 days up to 18 months in Part A of the study.
- PF-04360365 0.5 mg/kg (Part A): PF-04360365 0.5 mg/kg intravenous infusion over 2 hours every 60 days up to 18 months in Part A of the study.
- PF-04360365 1.0 mg/kg (Part A): PF-04360365 1.0 mg/kg intravenous infusion over 2 hours every 60 days up to 18 months in Part A of the study.
- Placebo (Part A): Placebo intravenous infusion over 2 hours every 60 days up to 18 months in Part A of the study.
- PF-04360365 3.0 mg/kg (Part B): PF-04360365 3.0 mg/kg intravenous infusion over 2 hours every 60 days up to 18 months in Part B of the study.
- PF-04360365 8.5 mg/kg (Part B): PF-04360365 8.5 mg/kg intravenous infusion over 2 hours every 60 days up to 18 months in Part B of the study.
- Placebo (Part B): Placebo intravenous infusion over 2 hours every 60 days up to 18 months in Part B of the study.
Period: Overall Study
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Started | 26 | 26 | 25 | 26 | 32 | 31 | 32
Treated | 25 | 25 | 25 | 24 | 32 | 31 | 32
Completed | 21 | 20 | 18 | 18 | 23 | 20 | 26
Not Completed | 5 | 6 | 7 | 8 | 9 | 11 | 6
Not completed — Adverse Event | 0 | 1 | 2 | 1 | 2 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 4 | 4 | 4 | 7 | 3
Not completed — Randomized, but not treated | 1 | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 1 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received an infusion of study medication (including partial infusions).
Groups:
- PF-04360365 0.1 mg/kg (Part A): PF-04360365 0.1 mg/kg intravenous infusion over 2 hours every 60 days up to 18 months in Part A of the study.
- Total: Total of all reporting groups
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B) | Total
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 32 | 31 | 32 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (8.2) | 71.9 (9.4) | 72.2 (8.4) | 70.0 (7.8) | 70.5 (8.9) | 71.8 (7.3) | 70.4 (10.3) | 71.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 11 | 13 | 20 | 17 | 17 | 105
  Male | 13 | 10 | 14 | 11 | 12 | 14 | 15 | 89

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. SAE: an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events between first dose of study medication and up to 6 months after last dose that were absent before treatment or worsened relative to pre-treatment state.
Time Frame: Day 1 up to 6 months after last dose of study medication, assessed up to Month 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 32 | 31 | 32
Participants
  AEs | 24 | 24 | 24 | 24 | 27 | 28 | 32
  SAEs | 7 | 8 | 7 | 3 | 7 | 10 | 3

2. Primary Outcome: Number of Participants With Change From Baseline in Brain Magnetic Resonance Imaging (MRI) Abnormalities
Description: Number of participants with new clinical findings not evident on the baseline scans, such as brain edema, hemorrhage, encephalitis and other pathology (cerebral/meningeal enhancement, parenchymal hematoma, subarachnoid hemorrhage, subdural hematoma, cortical infarcts, subcortical grey matter infarcts, white matter infarcts and white matter hyperintensities) were assessed from structural MRI. Participants with brain abnormality other than those listed above, assessed using MRI scan, were reported under other abnormality. Baseline was defined as the last assessment prior to the first study drug infusion.
Time Frame: Baseline up to Month 24
Population: Safety analysis set included all participants who received an infusion of study medication (including partial infusions). Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 31 | 28 | 32
Participants
  Cerebral Edema | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cerebral/Meningeal Enhancement | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Micro Hemorrhage | 4 | 7 | 2 | 6 | 3 | 6 | 6
  Subdural Hematoma | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Cortical Infarcts | 1 | 0 | 2 | 0 | 0 | 1 | 0
  Subcortical Grey Matter Infarcts | 0 | 0 | 0 | 0 | 1 | 1 | 0
  White Matter Infarcts | 0 | 1 | 0 | 0 | 0 | 0 | 2
  White Matter Hyper Intensities | 0 | 3 | 2 | 2 | 4 | 0 | 2
  Other Abnormality | 12 | 9 | 8 | 10 | 8 | 12 | 10

3. Primary Outcome: Number of Participants With Gadolinium Use in Brain Magnetic Resonance Imaging (MRI)
Description: Brain MRI included gadolinium contrast if investigator determined this was necessary for participant care either based on clinical signs or the non-contrast MRI. This decision was made by the investigator on the basis of change in the clinical examination or in response to a possible abnormality seen on the non-contrast brain MRI. Baseline was defined as the last assessment prior to the first study drug infusion.
Time Frame: Baseline up to Month 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 31 | 28 | 32
Participants | 3 | 1 | 2 | 1 | 1 | 2 | 3

4. Primary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of PF-04360365 at 0 Hour on Day 0
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour on Day 0
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 infusion of study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 3 | 8 | 4 | 13 | 11
Nanogram per milliliter | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)

5. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 1
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 1
Population: PK analysis set included all participants who received at least 1 infusion of study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 25 | 25 | 24 | 30 | 30
Nanogram per milliliter | 0.00 (0.00) | 0.00 (0.00) | 14.25 (69.81) | 0.00 (0.00) | 38.10 (208.68)

6. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 1
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 22 | 20 | 23 | 28 | 27
Nanogram per milliliter | 1731.36 (605.07) | 10051.85 (1857.36) | 21972.09 (6582.50) | 65832.36 (23334.31) | 187953.19 (36763.80)

7. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 60
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 60
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 29 | 29
Nanogram per milliliter | 33.96 (82.22) | 792.80 (217.31) | 1747.04 (311.05) | 6715.34 (3797.08) | 30517.76 (34018.99)

8. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 60
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 60
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 23 | 24 | 24 | 29 | 23
Nanogram per milliliter | 2018.13 (402.12) | 11372.46 (2730.02) | 23100.33 (5598.52) | 81464.62 (25466.75) | 209962.13 (64637.17)

9. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 on Day 90
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 90
Population: PK analysis set included all participants who received at least 1 infusion of study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 30 | 28
Nanogram per milliliter
  CSF: number analyzed (Participants) | 4 | 6 | 5 | 11 | 10
  CSF | 0.00 (0.00) | 0.00 (0.00) | 6.36 (14.22) | 43.44 (17.76) | 157.40 (85.17)
  Plasma | 286.20 (133.25) | 2074.48 (558.85) | 4277.88 (1073.25) | 16733.03 (5624.57) | 49141.68 (11941.83)

10. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 120
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 120
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 30 | 27
Nanogram per milliliter | 106.08 (116.00) | 1259.68 (360.11) | 2573.64 (622.86) | 8781.20 (3267.52) | 31916.04 (24631.87)

11. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 120
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 120
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 22 | 25 | 23 | 27 | 24
Nanogram per milliliter | 2083.14 (549.16) | 12229.60 (2813.13) | 25263.43 (6395.62) | 69437.52 (19262.08) | 191019.54 (65338.19)

12. Primary Outcome: Mean Plasma Concentration of PF-04360365 on Day 150
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 150
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 24 | 25 | 25 | 30 | 27
Nanogram per milliliter | 344.17 (157.08) | 2512.36 (804.43) | 4673.32 (932.48) | 17636.10 (6440.44) | 53918.22 (15265.59)

13. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 180
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 180
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 24 | 25 | 25 | 28 | 26
Nanogram per milliliter | 114.71 (137.86) | 1344.00 (556.59) | 2819.68 (819.68) | 9885.71 (3673.92) | 30306.81 (11823.33)

14. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 180
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 180
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 21 | 23 | 23 | 26 | 23
Nanogram per milliliter | 1959.05 (650.77) | 12096.22 (3346.68) | 24574.57 (5989.22) | 72597.58 (13930.48) | 194768.61 (42953.08)

15. Primary Outcome: Mean Plasma Concentration of PF-04360365 on Day 210
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 210
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 24 | 24 | 25 | 28 | 27
Nanogram per milliliter | 245.33 (233.16) | 2419.25 (1034.32) | 4935.00 (1349.38) | 17973.43 (6279.98) | 55881.07 (17445.49)

16. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 240
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 240
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 25 | 24 | 24 | 27 | 26
Nanogram per milliliter | 170.64 (389.00) | 1423.83 (582.13) | 2782.17 (1147.38) | 11221.22 (4030.07) | 31093.81 (11083.26)

17. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 240
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 240
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 21 | 22 | 24 | 25 | 23
Nanogram per milliliter | 1660.76 (511.32) | 10501.00 (2550.48) | 22340.46 (5364.94) | 80142.40 (15093.45) | 216585.87 (32947.73)

18. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 300
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 300
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 24 | 22 | 24 | 26 | 27
Nanogram per milliliter | 176.25 (140.95) | 1690.41 (1585.87) | 2958.13 (1150.02) | 11935.88 (3779.50) | 31766.30 (12335.11)

19. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 300
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 300
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 24 | 20 | 23 | 24 | 21
Nanogram per milliliter | 1919.42 (446.62) | 10774.35 (1736.85) | 22273.26 (6285.72) | 76511.29 (13832.35) | 207292.95 (50582.35)

20. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 360
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 360
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 23 | 21 | 23 | 26 | 23
Nanogram per milliliter | 247.52 (102.75) | 1377.95 (476.42) | 3161.00 (972.99) | 10643.58 (3986.99) | 31485.52 (12609.26)

21. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 360
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 360
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 22 | 19 | 21 | 24 | 19
Nanogram per milliliter | 2019.23 (396.63) | 11047.68 (2232.06) | 22833.43 (4544.54) | 71309.58 (12691.07) | 203124.84 (35756.46)

22. Primary Outcome: Mean Plasma Concentration of PF-04360365 on Day 390
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 390
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 22 | 21 | 22 | 26 | 23
Nanogram per milliliter | 411.00 (195.94) | 2344.76 (780.92) | 4902.36 (1373.05) | 18721.04 (6458.67) | 54956.65 (20091.21)

23. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 420
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 420
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 21 | 21 | 21 | 24 | 21
Nanogram per milliliter | 204.62 (123.72) | 1433.52 (550.12) | 3102.24 (1146.00) | 9711.42 (3012.62) | 30782.57 (11295.55)

24. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 420
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 420
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 18 | 19 | 18 | 21 | 16
Nanogram per milliliter | 1919.50 (600.41) | 11513.89 (1589.13) | 23519.67 (4499.54) | 69975.00 (16885.06) | 196647.81 (29248.03)

25. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 480
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 480
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 23 | 21 | 20 | 24 | 22
Nanogram per milliliter | 162.52 (161.33) | 1480.95 (557.75) | 3125.25 (1074.07) | 10585.67 (3272.66) | 26612.45 (12061.46)

26. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 480
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 480
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 21 | 19 | 19 | 21 | 18
Nanogram per milliliter | 1936.67 (484.01) | 11293.26 (2237.99) | 22930.21 (4146.48) | 67981.00 (10368.30) | 169955.72 (35843.29)

27. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 0 Hour on Day 540
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 0 Hour (pre-dose) on Day 540
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 23 | 19 | 16 | 23 | 23
Nanogram per milliliter | 177.30 (163.34) | 1297.26 (578.84) | 2718.38 (949.54) | 10372.65 (4310.28) | 32303.09 (35225.88)

28. Primary Outcome: Mean Plasma Concentration of PF-04360365 at 2 Hours on Day 540
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: 2 Hours on Day 540
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 20 | 15 | 15 | 22 | 18
Nanogram per milliliter | 1981.20 (591.23) | 11291.40 (2033.92) | 20793.73 (4168.51) | 70660.14 (16140.32) | 178273.50 (40289.00)

29. Primary Outcome: Mean Plasma and Cerebrospinal Fluid (CSF) Concentration of PF-04360365 on Day 570
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 570
Population: PK analysis set included all participants who received at least 1 infusion of study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified category for rows.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 22 | 21 | 18 | 22 | 22
Nanogram per milliliter
  CSF: number analyzed (Participants) | 2 | 4 | 3 | 10 | 7
  CSF | 0.00 (0.00) | 0.00 (0.00) | 6.30 (10.91) | 56.77 (23.14) | 115.36 (79.21)
  Plasma | 360.05 (165.65) | 2023.95 (911.00) | 4374.00 (1465.99) | 19638.68 (8134.26) | 44945.95 (25370.94)

30. Primary Outcome: Mean Plasma Concentration of PF-04360365 on Day 660
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 660
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 21 | 18 | 18 | 22 | 21
Nanogram per milliliter | 10.33 (47.35) | 480.78 (303.49) | 1212.22 (596.19) | 4196.50 (2342.84) | 7576.29 (5013.34)

31. Primary Outcome: Mean Plasma Concentration of PF-04360365 on Day 720
Description: Only participants received PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 720
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 21 | 20 | 18 | 23 | 20
Nanogram per milliliter | 0.00 (0.00) | 198.70 (206.30) | 590.56 (380.08) | 1583.22 (1163.66) | 2795.30 (1606.90)

32. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) Score at Baseline
Description: ADAS-cog is a structured scale assessing the severity of cognitive impairment in Alzheimer's Disease. It comprised of following 11 items (range): word recall (0-10), naming objects and fingers (0-5), following commands (0-5), constructional praxis (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), recall of test instructions (0-5), spoken language ability (0-5), word-finding difficulty (0-5), comprehension of spoken language (0-5). ADAS-cog total score was calculated as the sum of scores for the 11 items and ranged from 0 to 70. Higher total and individual item scores indicate greater cognitive impairment. Baseline was defined as the last assessment prior to the first study drug infusion.
Time Frame: Baseline
Population: Full analysis set (FAS) included all randomized participants who had received at least 1 infusion of study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 24 | 25 | 24 | 31 | 31 | 32
Units on a scale | 20.0 (7.87) | 20.4 (8.19) | 20.8 (6.08) | 20.0 (6.98) | 19.4 (6.96) | 24.5 (10.15) | 18.4 (7.45)

33. Secondary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) Score at Month 19
Description: as for outcome 32
Time Frame: Baseline and Month 19
Population: FAS included all randomized participants who had received at least 1 infusion of study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 22 | 18 | 16 | 18 | 21 | 21 | 27
Units on a scale | 8.36 (2.07) | 9.00 (2.20) | 9.25 (2.20) | 6.98 (2.22) | 9.58 (1.95) | 8.71 (1.99) | 7.85 (1.81)
Statistical Analysis 1: Comparison: PF-04360365 0.1 mg/kg (Part A) vs Placebo (Part A); Mixed model repeated measures used terms for treatment, visit, baseline value, country, and treatment-by-visit interaction, with unstructured covariance matrix; Test type: Superiority; p = 0.6504, Mixed Models Analysis; Least Squares (LS) Mean Difference = 1.38, 90% CI 2-sided [-3.68 to 6.45], Standard Error of Mean 3.04
Statistical Analysis 2: Comparison: PF-04360365 0.5 mg/kg (Part A) vs Placebo (Part A); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.5213, Mixed Models Analysis; LS Mean Difference = 2.02, 90% CI 2-sided [-3.20 to 7.23], Standard Error of Mean 3.13
Statistical Analysis 3: Comparison: PF-04360365 1.0 mg/kg (Part A) vs Placebo (Part A); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.4698, Mixed Models Analysis; LS Mean Difference = 2.27, 90% CI 2-sided [-2.94 to 7.48], Standard Error of Mean 3.13
Statistical Analysis 4: Comparison: PF-04360365 3.0 mg/kg (Part B) vs Placebo (Part B); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.5183, Mixed Models Analysis; LS Mean Difference = 1.73, 90% CI 2-sided [-2.71 to 6.17], Standard Error of Mean 2.66
Statistical Analysis 5: Comparison: PF-04360365 8.5 mg/kg (Part B) vs Placebo (Part B); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.7529, Mixed Models Analysis; LS Mean Difference = 0.85, 90% CI 2-sided [-3.65 to 5.35], Standard Error of Mean 2.70

34. Secondary Outcome: Disability Assessment for Dementia (DAD) Score at Baseline
Description: DAD is a functional assessment based on interview with the caregiver. It consisted of 40 items, 17 related to self-care and 23 items involving instrumental activities of daily living. Each item was scored as yes = 1, no = 0 and not applicable= N/A. A total score was obtained by adding the rating for each question and converting this to a total score out of 100. The items rated N/A were not considered for the total score. DAD total score ranged from 0 to 100, with higher scores indicating better functioning. Baseline was defined as the last assessment prior to the first study drug infusion.
Time Frame: Baseline
Population: FAS included all randomized participants who had received at least 1 infusion of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 32 | 31 | 32
Units on a scale | 79.6 (13.73) | 83.4 (12.83) | 78.1 (20.55) | 78.0 (16.40) | 83.5 (13.16) | 77.1 (20.16) | 80.7 (15.60)

35. Secondary Outcome: Change From Baseline in Disability Assessment for Dementia (DAD) Score at Month 19
Description: as for outcome 34
Time Frame: Baseline and Month 19
Population: as for outcome 33
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 21 | 21 | 18 | 18 | 24 | 22 | 27
Units on a scale | -20.09 (3.80) | -16.20 (3.90) | -15.18 (3.91) | -16.02 (4.07) | -22.53 (4.17) | -18.12 (4.30) | -18.44 (4.00)
Statistical Analysis 1: Comparison: PF-04360365 0.1 mg/kg (Part A) vs Placebo (Part A); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.4688, Mixed Models Analysis; LS Mean Difference = -4.07, 90% CI 2-sided [-13.38 to 5.24], Standard Error of Mean 5.59
Statistical Analysis 2: Comparison: PF-04360365 0.5 mg/kg (Part A) vs Placebo (Part A); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.9743, Mixed Models Analysis; LS Mean Difference = -0.18, 90% CI 2-sided [-9.59 to 9.22], Standard Error of Mean 5.64
Statistical Analysis 3: Comparison: PF-04360365 1.0 mg/kg (Part A) vs Placebo (Part A); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.8824, Mixed Models Analysis; LS Mean Difference = 0.84, 90% CI 2-sided [-8.57 to 10.25], Standard Error of Mean 5.65
Statistical Analysis 4: Comparison: PF-04360365 3.0 mg/kg (Part B) vs Placebo (Part B); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.4831, Mixed Models Analysis; LS Mean Difference = -4.09, 90% CI 2-sided [-13.77 to 5.58], Standard Error of Mean 5.81
Statistical Analysis 5: Comparison: PF-04360365 8.5 mg/kg (Part B) vs Placebo (Part B); [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.9562, Mixed Models Analysis; LS Mean Difference = 0.32, 90% CI 2-sided [-9.48 to 10.13], Standard Error of Mean 5.88

36. Secondary Outcome: Mean Plasma Concentration of Amyloid Beta 1-x (Aβ1-x)
Time Frame: 0 Hour (pre-dose) and 2 hours on Day 1, 60, 120, 180, 240, 300, 360, 420, 480, 540; Day 90, 150, 210, 390, 570, 660, 720
Population: FAS included all randomized participants who had received at least 1 infusion of study medication. Here 'Number Analyzed' signifies participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 32 | 31 | 32
Picogram per milliliter
  0 Hour Day 1: number analyzed (Participants) | 25 | 25 | 25 | 24 | 32 | 31 | 31
  0 Hour Day 1 | 294.12 (95.78) | 229.68 (112.23) | 355.80 (514.90) | 273.21 (96.00) | 607.50 (765.24) | 337.87 (112.84) | 382.10 (158.90)
  2 Hours Day 1: number analyzed (Participants) | 22 | 20 | 23 | 22 | 28 | 28 | 27
  2 Hours Day 1 | 2128.73 (537.63) | 2106.50 (480.76) | 2199.87 (621.29) | 282.86 (75.09) | 2446.64 (1055.11) | 2648.93 (695.78) | 380.07 (101.11)
  0 Hour Day 60: number analyzed (Participants) | 24 | 25 | 25 | 24 | 29 | 29 | 32
  0 Hour Day 60 | 1828.13 (976.47) | 8122.40 (2209.66) | 15558.40 (4994.54) | 332.46 (94.47) | 48603.45 (20147.32) | 91475.86 (22246.33) | 405.44 (245.46)
  2 Hours Day 60: number analyzed (Participants) | 23 | 23 | 24 | 21 | 29 | 22 | 29
  2 Hours Day 60 | 3892.17 (1013.64) | 9645.22 (1953.32) | 16952.50 (4358.13) | 291.62 (108.42) | 41772.41 (11979.65) | 83050.00 (28159.10) | 380.90 (119.24)
  Day 90: number analyzed (Participants) | 25 | 25 | 25 | 24 | 30 | 28 | 32
  Day 90 | 3997.20 (1322.48) | 20476.00 (5034.49) | 36904.00 (12258.21) | 341.33 (80.25) | 89856.67 (20377.45) | 127132.14 (25567.72) | 386.50 (167.65)
  0 Hour Day 120: number analyzed (Participants) | 25 | 24 | 25 | 23 | 30 | 27 | 32
  0 Hour Day 120 | 2440.00 (1054.77) | 11435.00 (3379.92) | 22416.00 (6636.56) | 340.87 (96.43) | 61270.00 (22462.23) | 110074.07 (23932.00) | 375.22 (118.27)
  2 Hours Day 120: number analyzed (Participants) | 22 | 25 | 23 | 20 | 27 | 23 | 29
  2 Hours Day 120 | 4425.05 (1427.10) | 12988.80 (4021.06) | 22260.87 (6276.85) | 361.80 (53.92) | 49233.33 (18308.66) | 91508.70 (20558.34) | 396.10 (117.46)
  Day 150: number analyzed (Participants) | 24 | 25 | 25 | 23 | 30 | 27 | 32
  Day 150 | 4531.25 (1597.31) | 23600.00 (6871.74) | 43872.00 (10714.22) | 360.30 (74.99) | 85203.33 (21436.55) | 135288.89 (29714.08) | 363.38 (126.56)
  0 Hour Day 180: number analyzed (Participants) | 24 | 25 | 25 | 22 | 28 | 25 | 31
  0 Hour Day 180 | 3017.50 (1296.78) | 14386.00 (5203.12) | 26036.00 (7745.58) | 367.55 (63.64) | 55125.00 (15273.79) | 93180.00 (28531.81) | 297.87 (122.91)
  2 Hours Day 180: number analyzed (Participants) | 21 | 23 | 22 | 18 | 25 | 23 | 29
  2 Hours Day 180 | 5544.76 (2044.34) | 16894.78 (5283.81) | 27118.18 (7787.09) | 363.61 (72.24) | 47316.00 (15189.79) | 81960.87 (26561.69) | 289.24 (139.31)
  Day 210: number analyzed (Participants) | 24 | 24 | 25 | 22 | 28 | 26 | 31
  Day 210 | 4673.33 (1524.00) | 25108.33 (8120.77) | 49676.00 (12637.16) | 385.27 (71.98) | 84810.71 (20382.91) | 116703.85 (37969.45) | 301.84 (110.90)
  0 Hour Day 240: number analyzed (Participants) | 25 | 24 | 24 | 21 | 27 | 26 | 30
  0 Hour Day 240 | 3085.20 (1190.23) | 15445.83 (5718.03) | 28520.83 (8766.83) | 327.29 (67.08) | 48344.44 (14065.65) | 83653.85 (28195.07) | 318.37 (116.19)
  2 Hours Day 240: number analyzed (Participants) | 21 | 22 | 24 | 21 | 25 | 24 | 29
  2 Hours Day 240 | 5269.05 (1614.58) | 15930.91 (6681.72) | 25532.50 (7102.35) | 336.24 (47.77) | 47100.00 (15547.48) | 78354.17 (28042.48) | 350.28 (130.39)
  0 Hour Day 300: number analyzed (Participants) | 25 | 22 | 24 | 21 | 26 | 27 | 30
  0 Hour Day 300 | 2963.6 (1047.13) | 14710.45 (6472.62) | 28366.67 (14592.96) | 311.43 (63.44) | 62607.69 (21254.16) | 96537.04 (44313.44) | 327.83 (112.77)
  2 Hours Day 300: number analyzed (Participants) | 24 | 20 | 23 | 20 | 24 | 21 | 29
  2 Hours Day 300 | 4984.58 (1496.74) | 15878.00 (7211.88) | 28647.83 (14306.10) | 297.20 (97.78) | 53808.33 (18101.79) | 79900.00 (26477.07) | 353.24 (129.21)
  0 Hour Day 360: number analyzed (Participants) | 23 | 21 | 23 | 21 | 26 | 23 | 28
  0 Hour Day 360 | 3053.04 (972.76) | 14313.81 (6254.35) | 27999.13 (13280.23) | 287.90 (103.73) | 58157.69 (15871.24) | 100691.30 (37696.25) | 353.86 (108.68)
  2 Hours Day 360: number analyzed (Participants) | 22 | 19 | 21 | 18 | 24 | 19 | 26
  2 Hours Day 360 | 5253.18 (1802.73) | 14153.16 (6473.23) | 23664.29 (11040.37) | 277.72 (94.14) | 50820.83 (16118.20) | 84168.42 (34779.51) | 351.31 (105.35)
  Day 390: number analyzed (Participants) | 22 | 21 | 22 | 21 | 26 | 23 | 28
  Day 390 | 4300.82 (1647.44) | 19984.76 (7108.94) | 40330.45 (13327.52) | 303.76 (125.67) | 75133.85 (23426.25) | 114104.35 (31087.60) | 338.79 (92.17)
  0 Hour Day 420: number analyzed (Participants) | 21 | 21 | 21 | 20 | 23 | 21 | 26
  0 Hour Day 420 | 3123.19 (1245.10) | 14675.24 (6367.51) | 26109.52 (13214.13) | 318.45 (76.39) | 55273.91 (22852.20) | 89038.10 (31754.61) | 376.08 (172.83)
  2 Hours Day 420: number analyzed (Participants) | 18 | 19 | 18 | 16 | 21 | 15 | 25
  2 Hours Day 420 | 5090.56 (1713.37) | 14711.58 (5023.57) | 23987.78 (9082.14) | 318.88 (61.86) | 54461.90 (22287.94) | 89080.00 (25517.79) | 394.04 (229.59)
  0 Hour Day 480: number analyzed (Participants) | 23 | 21 | 20 | 19 | 24 | 23 | 27
  0 Hour Day 480 | 2899.17 (1058.84) | 13864.29 (6772.94) | 29448.00 (11647.42) | 339.16 (86.94) | 75033.33 (29410.21) | 97239.57 (40197.50) | 356.11 (197.30)
  2 Hours Day 480: number analyzed (Participants) | 21 | 19 | 19 | 16 | 21 | 17 | 25
  2 Hours Day 480 | 5196.19 (1676.54) | 16105.79 (7332.47) | 28064.21 (11182.90) | 396.44 (98.10) | 77633.33 (35071.25) | 100941.18 (36351.53) | 402.72 (195.38)
  0 Hour Day 540: number analyzed (Participants) | 23 | 19 | 16 | 18 | 22 | 20 | 24
  0 Hour Day 540 | 3163.48 (1389.06) | 14449.47 (6474.26) | 32468.13 (14928.53) | 359.06 (91.66) | 53154.55 (18919.37) | 77400.00 (37951.50) | 493.71 (251.99)
  2 Hours Day 540: number analyzed (Participants) | 20 | 15 | 15 | 17 | 20 | 14 | 24
  2 Hours Day 540 | 5755.50 (3402.11) | 15516.00 (6002.06) | 30778.67 (16628.98) | 387.65 (119.66) | 54190.00 (20426.89) | 94271.43 (36384.07) | 455.04 (201.94)
  Day 570: number analyzed (Participants) | 22 | 21 | 17 | 17 | 21 | 21 | 24
  Day 570 | 4568.64 (2097.91) | 22257.14 (10734.97) | 49461.76 (22369.81) | 356.71 (151.05) | 69914.29 (19836.82) | 90576.19 (60817.37) | 400.58 (175.08)
  Day 660: number analyzed (Participants) | 21 | 18 | 18 | 17 | 22 | 21 | 26
  Day 660 | 2422.29 (1956.43) | 8181.11 (7497.62) | 20496.11 (20540.31) | 421.71 (140.09) | 28198.18 (10933.08) | 49011.19 (35384.55) | 475.46 (386.01)
  Day 720: number analyzed (Participants) | 21 | 20 | 18 | 18 | 23 | 20 | 25
  Day 720 | 1383.76 (449.57) | 3773.5 (2447.14) | 7876.67 (5846.23) | 419.11 (143.12) | 14912.65 (8037.28) | 22663.00 (14507.34) | 421.44 (170.96)

37. Secondary Outcome: Mean Plasma Concentration of Amyloid Beta 1-40 (Aβ1-40)
Time Frame: as for outcome 36
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 32 | 31 | 32
Picogram per milliliter
  0 Hour Day 1: number analyzed (Participants) | 25 | 25 | 25 | 24 | 32 | 31 | 31
  0 Hour Day 1 | 185.52 (109.70) | 145.92 (104.50) | 162.04 (125.00) | 180.54 (108.32) | 318.09 (495.37) | 192.03 (199.53) | 184.19 (124.59)
  2 Hours Day 1: number analyzed (Participants) | 22 | 20 | 23 | 22 | 28 | 28 | 27
  2 Hours Day 1 | 1239.41 (388.07) | 1580.70 (500.06) | 1665.57 (953.50) | 187.95 (55.99) | 1924.50 (773.00) | 1764.64 (546.77) | 180.22 (117.09)
  0 Hour Day 60: number analyzed (Participants) | 24 | 25 | 25 | 24 | 29 | 29 | 32
  0 Hour Day 60 | 1073.50 (409.71) | 5860.00 (1923.23) | 11643.20 (4588.36) | 209.46 (71.27) | 33203.45 (13116.74) | 66972.41 (19944.83) | 158.16 (121.12)
  2 Hours Day 60: number analyzed (Participants) | 23 | 23 | 24 | 21 | 29 | 22 | 29
  2 Hours Day 60 | 2502.39 (920.12) | 8676.09 (2600.95) | 14517.08 (6129.96) | 227.57 (60.84) | 32306.90 (11373.09) | 69627.27 (21824.67) | 195.83 (110.94)
  Day 90: number analyzed (Participants) | 25 | 25 | 25 | 24 | 30 | 28 | 32
  Day 90 | 2096.40 (896.20) | 13888.80 (5357.63) | 25008.00 (8167.92) | 204.25 (71.71) | 57333.33 (15829.03) | 95967.86 (27202.68) | 157.31 (107.72)
  0 Hour Day 120: number analyzed (Participants) | 25 | 24 | 25 | 23 | 30 | 27 | 32
  0 Hour Day 120 | 1345.72 (525.64) | 7823.75 (3119.88) | 16724.00 (7330.78) | 192.91 (110.77) | 36926.67 (15677.13) | 75514.81 (22013.70) | 168.41 (81.95)
  2 Hours Day 120: number analyzed (Participants) | 22 | 25 | 23 | 20 | 27 | 23 | 29
  2 Hours Day 120 | 3000.00 (1145.59) | 11108.00 (3594.09) | 20834.78 (8115.40) | 191.95 (76.36) | 38466.67 (12659.44) | 76860.87 (22351.34) | 177.55 (94.50)
  Day 150: number analyzed (Participants) | 24 | 25 | 25 | 23 | 30 | 27 | 32
  Day 150 | 2564.21 (1566.85) | 16254.80 (5774.43) | 27640.00 (11619.21) | 195.96 (78.74) | 52753.33 (19076.48) | 75033.33 (19112.32) | 148.47 (106.04)
  0 Hour Day 180: number analyzed (Participants) | 24 | 25 | 25 | 22 | 28 | 26 | 31
  0 Hour Day 180 | 1632.54 (931.22) | 8604.40 (3269.47) | 17727.60 (7878.69) | 182.41 (86.46) | 35539.29 (12873.73) | 67450.00 (21320.30) | 161.48 (166.60)
  2 Hours Day 180: number analyzed (Participants) | 21 | 23 | 22 | 18 | 25 | 23 | 29
  2 Hours Day 180 | 2973.05 (1614.36) | 11533.48 (3718.57) | 23146.36 (9074.15) | 225.17 (94.23) | 38644.00 (13630.61) | 61634.78 (21758.96) | 150.79 (99.12)
  Day 210: number analyzed (Participants) | 24 | 24 | 25 | 22 | 28 | 27 | 31
  Day 210 | 2274.58 (878.71) | 14409.58 (5966.02) | 28548.00 (11006.03) | 191.82 (92.92) | 51135.71 (14603.53) | 71200.00 (17902.92) | 189.13 (78.73)
  0 Hour Day 240: number analyzed (Participants) | 25 | 24 | 24 | 21 | 27 | 26 | 30
  0 Hour Day 240 | 1471.84 (549.70) | 8583.75 (4003.84) | 16937.08 (7343.63) | 164.29 (46.78) | 36451.85 (10133.13) | 58873.08 (21088.17) | 141.40 (106.52)
  2 Hours Day 240: number analyzed (Participants) | 21 | 22 | 24 | 21 | 25 | 24 | 29
  2 Hours Day 240 | 2868.10 (778.74) | 11830.45 (5542.51) | 20021.25 (7600.16) | 182.71 (60.37) | 35996.00 (9149.79) | 58225.00 (20401.28) | 171.66 (98.41)
  0 Hour Day 300: number analyzed (Participants) | 25 | 22 | 24 | 21 | 26 | 27 | 30
  0 Hour Day 300 | 1630.16 (662.16) | 8989.55 (4776.13) | 17817.08 (13181.85) | 190.38 (80.76) | 37692.31 (15132.16) | 55488.89 (17874.01) | 149.20 (122.88)
  2 Hours Day 300: number analyzed (Participants) | 24 | 20 | 23 | 20 | 24 | 21 | 29
  2 Hours Day 300 | 2756.25 (1012.41) | 10428.50 (2989.20) | 17809.57 (6105.73) | 208.85 (108.79) | 42245.83 (12637.11) | 54838.10 (14484.59) | 245.31 (239.90)
  0 Hour Day 360: number analyzed (Participants) | 23 | 21 | 23 | 21 | 26 | 23 | 28
  0 Hour Day 360 | 1694.26 (566.45) | 8194.76 (3665.29) | 15651.74 (5075.04) | 236.71 (190.38) | 30459.62 (13619.52) | 48904.35 (18386.82) | 87.18 (96.11)
  2 Hours Day 360: number analyzed (Participants) | 22 | 19 | 21 | 18 | 24 | 19 | 25
  2 Hours Day 360 | 3277.27 (983.77) | 11555.79 (3710.85) | 16970.95 (6137.24) | 211.33 (101.44) | 31191.67 (10742.40) | 64868.42 (30014.29) | 156.68 (148.86)
  Day 390: number analyzed (Participants) | 22 | 21 | 22 | 21 | 25 | 23 | 28
  Day 390 | 2543.50 (1446.05) | 10594.76 (3948.17) | 21660.45 (7216.95) | 150.81 (85.06) | 54165.20 (20804.90) | 77274.78 (33435.47) | 131.07 (102.02)
  0 Hour Day 420: number analyzed (Participants) | 21 | 21 | 21 | 20 | 24 | 21 | 26
  0 Hour Day 420 | 1451.33 (602.01) | 7863.81 (3449.31) | 14975.24 (7980.85) | 157.80 (91.81) | 47820.83 (23683.71) | 65819.05 (42467.11) | 201.31 (165.16)
  2 Hours Day 420: number analyzed (Participants) | 18 | 19 | 18 | 16 | 21 | 15 | 24
  2 Hours Day 420 | 2647.78 (826.97) | 10538.42 (4177.09) | 16612.22 (5658.05) | 151.13 (86.07) | 44047.62 (21069.28) | 70846.67 (41555.50) | 181.83 (123.40)
  0 Hour Day 480: number analyzed (Participants) | 23 | 21 | 20 | 18 | 23 | 22 | 25
  0 Hour Day 480 | 1931.78 (1339.28) | 10108.10 (5878.70) | 16535.00 (9242.28) | 139.61 (106.88) | 74334.78 (21163.94) | 77302.27 (44463.25) | 252.00 (135.67)
  2 Hours Day 480: number analyzed (Participants) | 21 | 19 | 19 | 15 | 21 | 18 | 23
  2 Hours Day 480 | 3336.29 (1529.23) | 12793.68 (5639.73) | 16610.00 (6540.14) | 133.53 (91.30) | 66049.05 (37625.89) | 102094.44 (43738.40) | 310.39 (302.75)
  0 Hour Day 540: number analyzed (Participants) | 23 | 19 | 16 | 18 | 22 | 21 | 23
  0 Hour Day 540 | 2437.70 (1483.48) | 10103.16 (6545.00) | 27048.75 (23150.54) | 190.94 (127.00) | 52720.91 (26005.06) | 77010.48 (50743.64) | 198.00 (114.84)
  2 Hours Day 540: number analyzed (Participants) | 20 | 15 | 15 | 16 | 20 | 16 | 23
  2 Hours Day 540 | 4149.30 (1711.36) | 12428.67 (6799.53) | 31972.67 (24882.62) | 186.69 (95.55) | 52960.00 (25018.95) | 84750.00 (42228.62) | 230.30 (71.67)
  Day 570: number analyzed (Participants) | 22 | 21 | 17 | 17 | 21 | 21 | 24
  Day 570 | 3147.27 (1910.78) | 16370.00 (10166.72) | 32728.24 (20157.92) | 237.12 (176.71) | 58548.10 (25034.67) | 77292.38 (46608.10) | 192.13 (104.14)
  Day 660: number analyzed (Participants) | 21 | 17 | 18 | 16 | 22 | 21 | 16
  Day 660 | 1318.67 (927.31) | 4411.24 (3426.58) | 8720.00 (4958.03) | 290.63 (244.94) | 27949.09 (14956.33) | 42087.62 (26245.07) | 321.46 (140.99)
  Day 720: number analyzed (Participants) | 21 | 20 | 17 | 18 | 23 | 20 | 25
  Day 720 | 913.57 (273.04) | 3631.50 (2062.26) | 6642.94 (5669.98) | 330.11 (112.78) | 13954.48 (9828.94) | 22094.00 (13058.87) | 358.04 (148.65)

38. Secondary Outcome: Mean Plasma Concentration of Amyloid Beta 1-42 (Aβ1-42)
Description: Results are not reported for PF-04360365 0.1, 0.5, 1.0 mg/kg, Placebo (Part A and B) arms because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
Time Frame: as for outcome 36
Population: FAS included all randomized participants who had received at least 1 infusion of study medication. Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 24 | 30 | 31 | 32
Picogram per milliliter
  0 Hour Day 1 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 picogram per milliliter [pg/mL]). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 13.43 (25.72) | 19.14 (46.75) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 1: number analyzed (Participants) | 25 | 25 | 25 | 24 | 25 | 28 | 32
  2 Hours Day 1 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 11.13 (24.15) | 22.23 (56.62) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 60: number analyzed (Participants) | 25 | 25 | 25 | 24 | 28 | 29 | 32
  0 Hour Day 60 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 24.82 (50.09) | 33.21 (51.41) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 60: number analyzed (Participants) | 25 | 25 | 25 | 24 | 29 | 22 | 32
  2 Hours Day 60 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 15.27 (38.72) | 60.77 (210.62) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  Day 90: number analyzed (Participants) | 25 | 25 | 25 | 24 | 27 | 28 | 32
  Day 90 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 15.34 (37.22) | 41.53 (89.72) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 120: number analyzed (Participants) | 25 | 25 | 25 | 24 | 30 | 27 | 32
  0 Hour Day 120 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 13.62 (31.54) | 32.26 (56.72) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 120: number analyzed (Participants) | 25 | 25 | 25 | 24 | 27 | 23 | 32
  2 Hours Day 120 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 11.35 (27.02) | 14.86 (37.79) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  Day 150: number analyzed (Participants) | 25 | 25 | 25 | 24 | 30 | 27 | 32
  Day 150 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 12.01 (32.98) | 43.57 (125.33) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 180: number analyzed (Participants) | 25 | 25 | 25 | 24 | 27 | 26 | 32
  0 Hour Day 180 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 13.11 (30.57) | 41.39 (77.77) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 180: number analyzed (Participants) | 25 | 25 | 25 | 24 | 25 | 23 | 32
  2 Hours Day 180 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 12.66 (27.27) | 21.64 (43.59) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  Day 210: number analyzed (Participants) | 25 | 25 | 25 | 24 | 27 | 27 | 32
  Day 210 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 10.08 (32.66) | 24.06 (57.43) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 240: number analyzed (Participants) | 25 | 25 | 25 | 24 | 27 | 26 | 32
  0 Hour Day 240 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 13.19 (26.27) | 35.47 (83.01) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 240: number analyzed (Participants) | 25 | 25 | 25 | 24 | 25 | 24 | 32
  2 Hours Day 240 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 8.83 (20.44) | 28.11 (66.93) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 300: number analyzed (Participants) | 25 | 25 | 25 | 24 | 26 | 27 | 32
  0 Hour Day 300 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 12.68 (25.00) | 55.96 (142.05) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 300: number analyzed (Participants) | 25 | 25 | 25 | 24 | 24 | 21 | 32
  2 Hours Day 300 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 12.21 (22.64) | 57.44 (156.63) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 360: number analyzed (Participants) | 25 | 25 | 25 | 24 | 26 | 23 | 32
  0 Hour Day 360 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 12.08 (30.02) | 66.16 (194.92) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 360: number analyzed (Participants) | 25 | 25 | 25 | 24 | 24 | 19 | 32
  2 Hours Day 360 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 11.93 (22.97) | 62.57 (164.16) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  Day 390: number analyzed (Participants) | 25 | 25 | 25 | 24 | 26 | 23 | 32
  Day 390 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 12.57 (30.68) | 72.92 (220.09) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 420: number analyzed (Participants) | 25 | 25 | 25 | 24 | 24 | 21 | 32
  0 Hour Day 420 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 9.89 (28.01) | 54.91 (131.76) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 420: number analyzed (Participants) | 25 | 25 | 25 | 24 | 21 | 15 | 32
  2 Hours Day 420 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 6.09 (22.85) | 64.51 (162.91) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 480: number analyzed (Participants) | 25 | 25 | 25 | 24 | 24 | 23 | 32
  0 Hour Day 480 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 6.94 (16.00) | 30.32 (91.79) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 480: number analyzed (Participants) | 25 | 25 | 25 | 24 | 21 | 18 | 32
  2 Hours Day 480 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 7.50 (14.00) | 37.13 (98.93) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  0 Hour Day 540: number analyzed (Participants) | 25 | 25 | 25 | 24 | 22 | 21 | 32
  0 Hour Day 540 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 5.05 (14.19) | 36.62 (87.98) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  2 Hours Day 540: number analyzed (Participants) | 25 | 25 | 25 | 24 | 20 | 16 | 32
  2 Hours Day 540 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 4.36 (11.09) | 26.73 (70.63) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  Day 570: number analyzed (Participants) | 25 | 25 | 25 | 24 | 21 | 21 | 32
  Day 570 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 4.53 (15.68) | 43.1 (114.46) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  Day 660: number analyzed (Participants) | 25 | 25 | 25 | 24 | 22 | 21 | 32
  Day 660 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 7.09 (33.26) | 26.21 (106.89) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).
  Day 720: number analyzed (Participants) | 25 | 25 | 25 | 24 | 22 | 19 | 32
  Day 720 | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL). | 7.70 (29.70) | 33.11 (144.30) | NA (NA) — Results are not reported because plasma Aβ1-42 concentrations were sporadic and below the lower limit of quantification (20 pg/mL).

39. Secondary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-x (Aβ1-x)
Time Frame: Day 0 (Hour 0), 90, 570
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 3 | 8 | 4 | 4 | 13 | 11 | 17
Picogram per milliliter
  Day 0 | 27400.00 (8361.22) | 30187.50 (10584.28) | 32150.00 (10033.44) | 18425.00 (5034.13) | 31553.85 (10242.12) | 25536.36 (9602.63) | 25923.53 (8724.93)
  Day 90: number analyzed (Participants) | 3 | 6 | 4 | 4 | 11 | 10 | 14
  Day 90 | 31766.67 (6906.04) | 31050.00 (9056.88) | 22775.00 (3856.06) | 16025.00 (3279.61) | 27850.00 (11601.40) | 31580.00 (16461.79) | 22888.57 (9294.70)
  Day 570: number analyzed (Participants) | 1 | 3 | 2 | 2 | 8 | 7 | 8
  Day 570 | 12200.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 32466.67 (7305.02) | 15250.00 (7424.62) | 11650.00 (1626.35) | 13378.75 (3643.53) | 10688.57 (2937.67) | 10467.50 (2876.30)

40. Secondary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-40 (Aβ1-40)
Time Frame: Day 0 (Hour 0), 90, 570
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 3 | 8 | 4 | 4 | 13 | 11 | 17
Picogram per milliliter
  Day 0 | 18100.00 (4513.31) | 11907.50 (3569.78) | 11700.00 (1525.34) | 7947.50 (2501.00) | 14672.31 (6776.14) | 12301.82 (4272.94) | 12713.53 (5960.78)
  Day 90: number analyzed (Participants) | 3 | 6 | 4 | 4 | 11 | 10 | 14
  Day 90 | 16833.33 (4244.21) | 14733.33 (4341.27) | 12350.00 (2537.06) | 7977.50 (1542.95) | 14106.36 (5225.42) | 13733.00 (4712.08) | 11745.71 (3627.05)
  Day 570: number analyzed (Participants) | 1 | 4 | 2 | 2 | 9 | 6 | 8
  Day 570 | 4930.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 10775.00 (5811.55) | 8445.00 (2128.39) | 5235.00 (572.76) | 7108.89 (1712.55) | 9315.00 (3779.86) | 4730.00 (1235.86)

41. Secondary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Amyloid Beta 1-42 (Aβ1-42)
Time Frame: Day 0 (Hour 0), 90, 570
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 3 | 8 | 4 | 4 | 13 | 11 | 17
Picogram per milliliter
  Day 0 | 983.00 (370.31) | 800.13 (267.63) | 851.75 (17.75) | 694.00 (217.22) | 959.54 (281.30) | 817.36 (323.31) | 803.41 (232.38)
  Day 90: number analyzed (Participants) | 3 | 6 | 4 | 4 | 11 | 10 | 14
  Day 90 | 1009.00 (298.29) | 821.33 (235.97) | 866.00 (176.40) | 557.50 (159.32) | 949.36 (223.50) | 895.80 (273.28) | 778.29 (221.01)
  Day 570: number analyzed (Participants) | 1 | 3 | 1 | 2 | 9 | 6 | 8
  Day 570 | 802.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 803.00 (7.55) | 958.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 421.50 (142.13) | 487.11 (483.28) | 582.33 (489.19) | 665.25 (358.57)

42. Secondary Outcome: Mean Cerebrospinal Fluid (CSF) Concentration of Total Tau and Phospho-tau (P-tau)
Time Frame: Day 0 (Hour 0), 90, 570
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 3 | 8 | 4 | 4 | 13 | 11 | 17
Picogram per milliliter
  Day 0: tau | 188.90 (118.60) | 223.79 (99.03) | 190.43 (102.86) | 96.13 (34.73) | 219.09 (192.54) | 167.40 (101.42) | 196.31 (147.04)
  Day 90: tau: number analyzed (Participants) | 3 | 6 | 4 | 4 | 10 | 10 | 13
  Day 90: tau | 202.33 (112.51) | 210.33 (98.42) | 167.78 (83.20) | 117.38 (22.52) | 217.64 (149.25) | 169.76 (121.25) | 158.00 (62.91)
  Day 570: tau: number analyzed (Participants) | 1 | 4 | 2 | 2 | 8 | 7 | 8
  Day 570: tau | 78.00 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 158.98 (93.46) | 90.80 (28.57) | 49.20 (5.37) | 166.18 (115.72) | 139.94 (83.16) | 124.24 (51.28)
  Day 0: p-tau | 72.53 (10.46) | 65.89 (28.22) | 49.13 (13.83) | 34.98 (11.40) | 56.72 (30.64) | 49.45 (23.76) | 59.17 (28.41)
  Day 90: p-tau: number analyzed (Participants) | 3 | 6 | 4 | 3 | 10 | 10 | 13
  Day 90: p-tau | 73.27 (7.28) | 70.15 (31.21) | 64.50 (30.38) | 47.13 (19.96) | 60.26 (36.98) | 57.77 (31.63) | 47.98 (16.91)
  Day 570: p-tau: number analyzed (Participants) | 1 | 4 | 2 | 2 | 8 | 7 | 8
  Day 570: p-tau | 70.70 (NA) — Standard deviation was not estimable since only 1 participant was evaluable. | 112.10 (45.51) | 76.45 (50.28) | 53.65 (34.58) | 54.43 (31.79) | 42.47 (16.69) | 53.59 (32.04)

43. Secondary Outcome: Number of Participants With Abnormal Cerebrospinal Fluid (CSF) Protein, Red Blood Cells (RBCs), White Blood Cells (WBCs), and Glucose Concentration
Description: Abnormality was defined as concentration either less than lower limit of normal (LLN) or more than upper limit of normal (ULN). Baseline was defined as the last assessment prior to the first study drug infusion
Time Frame: Baseline up to Month 24
Population: Safety analysis set included all participants who received an infusion of study medication (including partial infusions). Here "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Number analyzed (Participants) | 4 | 6 | 5 | 5 | 11 | 10 | 14
Participants
  CSF Protein (>ULN) | 1 | 3 | 1 | 3 | 4 | 4 | 4
  CSF RBCs (>ULN): number analyzed (Participants) | 4 | 6 | 5 | 5 | 10 | 9 | 11
  CSF RBCs (>ULN) | 2 | 2 | 4 | 1 | 6 | 2 | 5
  CSF WBCs (>ULN): number analyzed (Participants) | 4 | 6 | 5 | 5 | 11 | 9 | 14
  CSF WBCs (>ULN) | 0 | 0 | 0 | 0 | 2 | 0 | 0
  CSF Glucose (>ULN) | 2 | 0 | 0 | 0 | 2 | 2 | 3

44. Secondary Outcome: Number of Participants With Serum Anti-Drug Anti Body (ADA)
Description: Serum samples were analyzed for the presence or absence of anti-PF-04360365 antibodies using validated semi-quantitative enzyme linked immunosorbent assay (ELISA). Only participants receiving PF-04360365 were analyzed for this outcome measure.
Time Frame: Day 1 up to Month 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B)
Number analyzed (Participants) | 25 | 25 | 25 | 32 | 31
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-04360365 0.1 mg/kg (Part A) | PF-04360365 0.5 mg/kg (Part A) | PF-04360365 1.0 mg/kg (Part A) | Placebo (Part A) | PF-04360365 3.0 mg/kg (Part B) | PF-04360365 8.5 mg/kg (Part B) | Placebo (Part B)
Serious Adverse Events (participants affected / at risk) | 7/25 | 8/25 | 7/25 | 3/24 | 7/32 | 10/31 | 3/32
Other Adverse Events (participants affected / at risk) | 24/25 | 24/25 | 23/25 | 24/24 | 26/32 | 28/31 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04360365 0.1 mg/kg (Part A) (N=25) | PF-04360365 0.5 mg/kg (Part A) (N=25) | PF-04360365 1.0 mg/kg (Part A) (N=25) | Placebo (Part A) (N=24) | PF-04360365 3.0 mg/kg (Part B) (N=32) | PF-04360365 8.5 mg/kg (Part B) (N=31) | Placebo (Part B) (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrong drug administered (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Meningeal disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural hygroma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04360365 0.1 mg/kg (Part A) (N=25) | PF-04360365 0.5 mg/kg (Part A) (N=25) | PF-04360365 1.0 mg/kg (Part A) (N=25) | Placebo (Part A) (N=24) | PF-04360365 3.0 mg/kg (Part B) (N=32) | PF-04360365 8.5 mg/kg (Part B) (N=31) | Placebo (Part B) (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0 | 0 | 1 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid retraction (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pupils unequal (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 1 | 2 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 3 | 3 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 5 | 1 | 2 | 1 | 5
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 3 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis atrophic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 1 | 1 | 4 | 3 | 1
Palatal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 4 | 1 | 0 | 0 | 0 | 3
Asthenia (General disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 0
Fatigue (General disorders) | 4 | 3 | 5 | 1 | 4 | 4 | 3
Gait disturbance (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 2 | 0 | 3 | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 2 | 2 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 2
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 4 | 0 | 2 | 1 | 5 | 3 | 4
Onychomycosis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 0 | 1 | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 5 | 7 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 4 | 3 | 2 | 3 | 4 | 2 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bladder injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 4 | 1 | 2 | 6 | 2 | 5
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 3 | 3 | 8 | 4 | 9
Foreign body (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gas poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 3 | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 4 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nail injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bleeding time prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose fluctuation (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 2 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Carotid bruit (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatic specific antigen abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin B12 increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 3 | 4 | 1 | 2 | 3 | 1
Weight increased (Investigations) | 4 | 2 | 1 | 2 | 2 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 1 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haemosiderosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 3 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 1 | 3 | 2 | 4
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 1 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 0 | 1 | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bradykinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain stem microhaemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Cerebellar microhaemorrhage (Nervous system disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 0
Cerebral atrophy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cerebral microhaemorrhage (Nervous system disorders) | 4 | 6 | 1 | 6 | 2 | 6 | 5
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chorea (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cogwheel rigidity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 3 | 3 | 1 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspraxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gait apraxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 1 | 4 | 6 | 5 | 8
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperreflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intention tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pleurothotonus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2
Subdural hygroma (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Superficial siderosis of central nervous system (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 2 | 0
Upper motor neurone lesion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 2 | 2 | 1 | 1 | 1 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 4 | 3 | 3 | 2 | 4 | 2
Anxiety (Psychiatric disorders) | 3 | 5 | 1 | 3 | 3 | 3 | 2
Apathy (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 1 | 3 | 6 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 4 | 0 | 0 | 2 | 3
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Disinhibition (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 3 | 4 | 2 | 0
Jealous delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Paranoia (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Sleep talking (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stereotypy (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atonic urinary bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enuresis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 2 | 0 | 1 | 2 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 1 | 1 | 0 | 2 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 2 | 1 | 1 | 1 | 2 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 4 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 8 | 4 | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 1 | 1 | 1 | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 2 | 2
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menopause (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Verbal abuse (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic disorder (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2
Haematoma (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 3 | 0 | 1 | 4 | 1 | 2
Hypotension (Vascular disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0
Infarction (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Data for CSF protein, RBCs, WBCs, and glucose was recorded as number of participants with laboratory test abnormalities and not as change from baseline values as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.